CLINICAL TRIAL: NCT06678542
Title: A Phase 1, Open-label, Single-site, Randomized, Single-dose, Two-Period, Crossover Study to Assess the Relative Bioavailability of GP681 Powder for Oral Suspension and Tablet Formulations in Healthy Chinese Male Subjects
Brief Title: Study to Assess Relative Bioavailability of GP681 Formulations in Healthy Chinese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024-GP681-S-BA/CRC-C2413
Record Dates: First submitted 2024-10-30; First posted 2024-11-07 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Suspensions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment sequence T-R (Experimental)
  Interventions: Drug: GP681 tablet; Drug: GP681 Powder for Oral Suspension
- Treatment sequence R-T (Experimental)
  Interventions: Drug: GP681 tablet; Drug: GP681 Powder for Oral Suspension

INTERVENTIONS:
Drug: GP681 tablet — GP681 tablet, 20 mg, single oral dose in each Group.
  Other Names: Reference treatment
Drug: GP681 Powder for Oral Suspension — GP681 Powder for Oral Suspension, 20 mg, single oral dose in each Group.
  Other Names: Test Treatment

SUMMARY:
The primary objective is to evaluate the relative bioavailability and pharmacokinetic profile of a single oral dose of the test formulation, GP681 Powder for Oral Suspension (20 mg/sachet), compared to the reference formulation, GP681 tablet (20 mg/tablet), in healthy Chinese male subjects. The secondary objectives are to assess the safety of a single oral dose of the GP681 Powder for Oral Suspension (20 mg/sachet) and GP681 tablet (20 mg/tablet) in healthy Chinese male subjects, as well as the palatability (taste acceptability) of the GP681 Powder for Oral Suspension.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: Healthy male subjects.
2. Age: 18 to 45 years (inclusive).
3. Body Weight: Body mass index (BMI = weight (kg)/height2 (m2)) between 19.0 and 26.0 kg/m2 (inclusive), with body weight ≥ 50.0 kg.
4. Taste Perception Ability: Successfully passed the taste perception ability test.
5. Informed Consent: Fully understands the study's purpose, nature, requirements, methodology, and potential adverse reactions; voluntarily agrees to participate in the clinical trial and signs the informed consent form prior to any study procedures.
6. Contraception: Subject (and their partner) has no plans to conceive or donate sperm from the time of first dosing until 3 months after the last dose and agrees to use effective contraception during this period.

Exclusion Criteria:

1. Clinically significant abnormalities, as determined by the investigator, including history of neurological, respiratory, cardiovascular, gastrointestinal, urinary, hematological and lymphatic, endocrine, musculoskeletal, or other disorders that could affect study results, or history of gastrointestinal disease within 3 months prior to screening.
2. Inability to accurately express true taste perception.
3. Dysfunction in taste or olfactory senses.
4. Known hypersensitivity or allergy to the investigational product or any of its components (e.g., copovidone, crospovidone, lactose, microcrystalline cellulose, mannitol, maltitol, hydroxypropyl methylcellulose, colloidal silicon dioxide, sodium stearyl fumarate, sucralose, strawberry flavoring), or history of allergic diseases or a predisposition to allergies.
5. Clinically significant abnormalities in vital signs, physical examination, clinical laboratory tests, 12-lead ECG, or chest X-ray (posteroanterior view), or QTcF >450 ms, as assessed by the investigator.
6. Positive test results for hepatitis B surface antigen (HBsAg), HCV antibodies, Treponema pallidum antibodies, or HIV antibodies.
7. Smoking ≥10 cigarettes per day within 3 months prior to the first dose.
8. Surgical procedure within 3 months before the first dose or planned surgery during the study period.
9. Blood donation or significant blood loss ≥400 mL within 3 months before the first dose, or plans to donate blood within 3 months after the study.
10. Participation in another clinical drug trial within 3 months before the first dose.
11. Difficulty swallowing.
12. Intolerance to skin puncture, fear of blood or needles, or poor venous access for blood sampling.
13. Special dietary requirements or inability to adhere to the provided diet and study dietary restrictions.
14. Positive urine drug screen, history of substance abuse within the past 5 years, or use of illicit drugs within 3 months before the first dose.
15. Alcohol consumption exceeding 21 units per week (1 unit = 360 mL beer, 45 mL spirits with 40% alcohol, or 150 mL wine) within 6 months prior to screening, or a positive breath alcohol test.
16. Use of any drugs known to inhibit or induce hepatic drug metabolism (e.g., inducers like barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; inhibitors like SSRIs, cimetidine, diltiazem, macrolides, nitroimidazoles, sedatives, verapamil, fluoroquinolones, antihistamines) within 30 days before the first dose.
17. Use of any prescription drugs, over-the-counter medications, herbal remedies, or supplements within 2 weeks prior to the first dose.
18. Vaccination within 2 weeks before the first dose, or planned vaccination during the study.
19. Consumption of foods or beverages rich in caffeine, poppy seeds, and/or theobromine, theophylline, or grapefruit (e.g., coffee, strong tea, chocolate, caffeinated carbonated drinks, cola, grapefruit juice) within 48 hours before the first dose, or engaging in vigorous exercise within 48 hours before the first dose.
20. Any other condition deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-02-16 (Actual); Study Completion 2025-02-16 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 360 hours post-dose
Area under the plasma concentration-time curve from time zero to time of the last quantifiable concentration[AUC(0-T)] | Up to 360 hours post-dose
Area under the plasma concentration-time curve from time zero extrapolated to infinite time[AUC(INF)] | Up to 360 hours post-dose

SECONDARY OUTCOMES:
Time of maximum observed concentration(Tmax) | Up to 360 hours post-dose
Apparent terminal half-life (T-HALF) | Up to 360 hours post-dose
Incidence of adverse events (AEs) | Up to approximately 1 month post-dose
Incidence of serious adverse events (SAEs) | Up to approximately 1 month post-dose
Incidence of participants with vital sign abnormalities | Up to approximately 1 month post-dose
Incidence of participants with physical examinations abnormalities | Up to approximately 1 month post-dose
Incidence of participants with electrocardiogram (ECG) abnormalities | Up to approximately 1 month post-dose
Incidence of participants with clinical laboratory abnormalities | Up to approximately 1 month post-dose
Palatability Evaluation | Up to 24 hours post-dose
  The palatability of GP681 Powder for Oral Suspension will be evaluated to characterize and quantify the sensory attributes of the product, such as basic tastes (including bitterness, astringency, sweetness) and texture (grittiness). Overall acceptability will also be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Women and Children's hospital of Ningbo University, Ningbo, China

IPD SHARING:
Plan to Share IPD: No